CLINICAL TRIAL: NCT00202709
Title: Can Thought Field Therapy (TFT) be Helpful for Patients With an Anxiety Disorder, a Prospective, Randomized Pilot Study With Wait List as Control Group.
Brief Title: Can Thought Field Therapy (TFT) be Helpful for Patients With an Anxiety Disorder?
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sorlandet Hospital HF (Other Government)
Responsible Party: Audun Irgens, MD, Sorlandet sykehus HF
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SSHF-AUIR-1
Record Dates: First submitted 2005-09-12; First posted 2005-09-20 (Estimated); Last update posted 2011-07-28 (Estimated); Status verified 2005-09

CONDITIONS: Agoraphobia; Social Phobia; PTSD
Keywords: Anxiety disorder; Thought Field Therapy; Psychotherapy; Agoraphobia; Social Phobia; Post Traumatic Stress Disorder
MeSH Terms: conditions — Agoraphobia; Phobia, Social; Stress Disorders, Post-Traumatic; Anxiety Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Thought Field Therapy (TFT) (Experimental): Treatment with TFT, first one hour, then 1/2 hour.
  Interventions: Behavioral: Thought Field Therapy (TFT)
- Wait list control (No Intervention)

INTERVENTIONS:
Behavioral: Thought Field Therapy (TFT) — Treatment with TFT twice in one week
  Other Names: Wait list control
  Arms: Thought Field Therapy (TFT)

SUMMARY:
The purpose of this study is to find out if Thought Field Therapy has effect on certain anxiety disorders; agoraphobia, social phobia, and post traumatic stress disorder (PTSD).

DETAILED DESCRIPTION:
Thought Field Therapy is an alternative treatment method that has been shown, by casuistic reports, to give good results when applied for anxiety disorders. In this study 52 patients, with one or more of the diagnoses agoraphobia, social phobia and/or PTSD, where randomized to either treatment with TFT or a wait list. The treatment group all got treatment in one week. 2 1/2 months later both the treatment group and the control group were tested on the same items as before the treatment started. After this evaluation phase the control group got the same treatment as the treatment or study group. Both groups were evaluated 3 and 12 months after treatment, the study group also 6 months after treatment. 4 patients were omitted because they changed groups. The study were performed from May 2002 until June 2003.

ELIGIBILITY:
Inclusion Criteria:

* One or more of the study diagnoses agoraphobia, social phobia and/or PTSD

Exclusion Criteria:

* Ongoing psychosis
* Ongoing serious drug problems

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 52 (Actual)
Dates: Start 2002-05; Primary Completion 2003-08 (Actual); Study Completion 2003-08 (Actual)

PRIMARY OUTCOMES:
Global symptom index (gsi) on the Symptom checklist 90 revised (SCL-90-R) | Before treatment/wait list period, just after treatment, 3 months and 12 months after treatment. Group A also 6 months after treatment.

SECONDARY OUTCOMES:
Davidson Trauma Scale | Before treatment/wait list period, just after treatment, 3 months and 12 months after treatment. Group A also 6 months after treatment.
Liebowitz Social Anxiety Scale | Before treatment/wait list period, just after treatment, 3 months and 12 months after treatment. Group A also 6 months after treatment.
Hospital Anxiety and Depression Scale (HADS) | Before treatment/wait list period, just after treatment, 3 months and 12 months after treatment. Group A also 6 months after treatment.
Fear Questionnaire (FQ) | Before treatment/wait list period, just after treatment, 3 months and 12 months after treatment. Group A also 6 months after treatment.
Sheehan Disability Scale | Before treatment/wait list period, just after treatment, 3 months and 12 months after treatment. Group A also 6 months after treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Audun C Irgens, MD, Principal Investigator — Sorlandet Hospital HF
Locations (1):
- Sorlandet Hospital, Arendal, Norway

REFERENCES:
- [Derived] Irgens A, Dammen T, Nysaeter TE, Hoffart A. Thought Field Therapy (TFT) as a treatment for anxiety symptoms: a randomized controlled trial. Explore (NY). 2012 Nov-Dec;8(6):331-8. doi: 10.1016/j.explore.2012.08.002. PMID 23141789